CLINICAL TRIAL: NCT01367067
Title: Prediction of Claustrophobia During MR Imaging: An Observational 18-Months Single Center Study
Brief Title: Prediction of Claustrophobia During MR Imaging
Acronym: CLAUSTRO II
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marc Dewey, Professor of Radiology, Charite University, Berlin, Germany
Other Study IDs: EA1/020/08/E
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Claustrophobia
Keywords: claustrophobia; magnetic resonance imaging; MRI; anxiety; anxious patients; phobic disorders; anxiety disorders; mental disorders
MeSH Terms: conditions — Claustrophobia; Anxiety Disorders; Phobic Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Psychometric Questionnaire: Adult inpatients and outpatients with a clinical indication of any part of the body who have been referred to Charité for MR imaging and have filled out a psychometric questionnaire
- No Psychometric Questionnaire: Adult inpatients and outpatients with a clinical indication of any part of the body who have been referred to Charité for MR imaging and did not fill out a psychometric questionnaire

SUMMARY:
The objective of the study is to search for possible predictors for claustrophobia during magnetic resonance (MR) imaging. A claustrophobic event shall be defined by an incomplete examination, or a complete examination that requires coping actions by the staff. Coping actions may consist of the administration of sedatives, prism glasses, an MR imaging test run with the patient, a pause, the prone position, an escort in the scanner room, and supportive communication. The investigators hypothesize that there is a difference between patients with and without events in their scores on the Claustrophobia Questionnaire and several further psychometric questions. Other factors may also favour events like patient characteristics, examined region, duration of the examination and scanner type. Therefore, predictors could identify patients who are likely to experience claustrophobia during MR imaging so that they can receive the appropriate support by the staff to complete their examination. Thus a larger patient population could benefit from MR imaging.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients referred to MR imaging with a clinical indication of any part of the body
* Mentally and physically able to fill out a questionnaire
* Sufficient German language skills

Exclusion Criteria:

* Age under 18 years
* Patients from the Intensive Care Unit
* Severe emergencies
* Surgery during MR imaging
* Participation in other studies
* Fetal and prenatal examinations
* Referral from medical jurisprudence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult inpatients and outpatients with a clinical indication of any part of the body who are referred to Charité for MR imaging
Sampling Method: Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The mean score of the Claustrophobia Questionnaire for the prediction of a claustrophobic event during MR imaging | Up to 5 min after the end of the MR

SECONDARY OUTCOMES:
Identification of specific psychometric questions for the prediction of a claustrophobic event during MR imaging | Up to 5 min after the end of the MR
Identification of influential factors for the prediction of a claustrophobic event | Up to 5 min after the end of the MR

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, PD Dr. med., Principal Investigator — Charité
Locations (1):
- Charité, Berlin, Germany

REFERENCES:
- [Background] Dewey M, Schink T, Dewey CF. Claustrophobia during magnetic resonance imaging: cohort study in over 55,000 patients. J Magn Reson Imaging. 2007 Nov;26(5):1322-7. doi: 10.1002/jmri.21147. PMID 17969166
- [Background] Dewey M, Schink T, Dewey CF. Frequency of referral of patients with safety-related contraindications to magnetic resonance imaging. Eur J Radiol. 2007 Jul;63(1):124-7. doi: 10.1016/j.ejrad.2007.01.025. Epub 2007 Mar 23. PMID 17383136
- [Background] Enders J, Zimmermann E, Rief M, Martus P, Klingebiel R, Asbach P, Klessen C, Diederichs G, Bengner T, Teichgraber U, Hamm B, Dewey M. Reduction of claustrophobia during magnetic resonance imaging: methods and design of the "CLAUSTRO" randomized controlled trial. BMC Med Imaging. 2011 Feb 10;11:4. doi: 10.1186/1471-2342-11-4. PMID 21310075
- [Result] Napp AE, Enders J, Roehle R, Diederichs G, Rief M, Zimmermann E, Martus P, Dewey M. Analysis and Prediction of Claustrophobia during MR Imaging with the Claustrophobia Questionnaire: An Observational Prospective 18-month Single-Center Study of 6500 Patients. Radiology. 2017 Apr;283(1):148-157. doi: 10.1148/radiol.2016160476. Epub 2016 Nov 25. PMID 27892781
- See also: Radiology at Charité — http://radiologie.charite.de/